CLINICAL TRIAL: NCT04873128
Title: Comparative Genetic and Immune Response Analysis of Different COVID-19 Vaccine Candidates Using Multi-OMICS Approach
Acronym: COVID 19-VAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COVID 19-VAC
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Genetic Predisposition
Keywords: Multi-OMICS; COVID-19; Side effect; Immun response; Vaccination; Memory response
MeSH Terms: conditions — Genetic Predisposition to Disease; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy adults (Experimental): Healthy adults who had no infection with SARS-CoV-2 virus before or had recovered from COVID-19 and plan to take the various COVID-19 experimental vaccine candidates or had already one dose of COVID-19 vaccine and are going to have the second vaccination with a different vaccine.
  Study related procedures:
  1-3 days before application of the first vaccine dose (blood sample 1) 7-10 days after first dose of vaccine (blood sample 2), 1-3 days before second dose of vaccine (blood sample 3) 7-10 days after second vaccine dose (blood sample 4) 6-12 Months after second vaccine dose (blood sample 5, optional) Next Generation Sequencing (NGS) analysis and other omics analysis (transcriptomics, proteomics, metabolomics).
  Interventions: Genetic: Multi-OMICS
- COVID-19 vaccinated subjects with side effects (Experimental): COVID-19 vaccinated subjects with diagnosed central thrombosis, anaphylactic shock or other major or minor complications such as dermatitis.
  Study related procedures: Blood sample will be taken without time frame 1-3 days after admission to the hospital (severe side effects) or consulting a doctor (mild side effects) (blood sample 1) during treatment (blood sample 2) After subject is recovered (blood sample 3) 6-12 Months after recovering (blood sample 4, optional) Next Generation Sequencing (NGS) analysis and other omics analysis (transcriptomics, proteomics, metabolomics).
  Interventions: Genetic: Multi-OMICS

INTERVENTIONS:
Genetic: Multi-OMICS — Measurement of gene expression in immune cells (Human Peripheral Blood Mononuclear Cell (PBMCs) or total blood) using functional genomics, proteomics, metabolomics and lipidomics tools and compare the dynamics of immune response before and after vaccination against COVID-19.

SUMMARY:
Reaction of the immune system and the body to a Coronavirus-19 (COVID-19) vaccination is so different and ultimately unpredictable has not yet been clarified. It is also not yet known why people who have been vaccinated react to a vaccination with sometimes serious side effects. Using high-throughput dissecting (analytical) methods with the suffix OMICS ("Multi-OMICS" methods, collective characterization and quantification of pools of biological molecules) used in this study on the basis of blood tests, data from several molecular levels can be recorded and a holistic picture can be created from this, which can depict the connections between these levels.

DETAILED DESCRIPTION:
Various vaccines against COVID-19 ("CORONA") have now been approved in Germany. How and why the reaction of the immune system and the body to a COVID-19 vaccination is so different and ultimately unpredictable has not yet been clarified. It is also not yet known why people who have been vaccinated react to a vaccination with sometimes serious side effects. There are now initial indications that genetic prerequisites can play a role in the development of the immune response. Furthermore, we want to examine the long-term protection against Severe Acute Respiratory Syndrome Coronavirus Type 2 (SARS-CoV-2) infection through vaccination and learn to understand it better.

Using high-throughput dissecting (analytical) methods with the suffix OMICS ("Multi-OMICS" method) used in this study on the basis of blood tests, data from several molecular levels can be recorded and a holistic picture can be created from this, which can depict the connections between these levels.

The expected results can help to gain a better understanding of the underlying reactions to a COVID-19 vaccination and the functioning of the body (pathophysiology) in the future, which could enable the basis for the development of causal therapeutic approaches and improved vaccines.

ELIGIBILITY:
Inclusion Criteria:

Group 1

* Healthy donors (HD) who had recovered from COVID-19 disease and/or HD who did not have COVID-19 disease in the past
* and who will receive the COVID-19 vaccine or a COVID19 vaccine candidate or other protective vaccines
* HD who did receive one dose of a specific COVID19 vaccine but who will receive a different vac-cine for her/his second vaccination for completion of the immunization
* Age > 18 years

Group 2

* Vaccinated subjects who are diagnosed with central thrombosis, anaphylactic shock or other major or minor complications such as atopic dermatitis (for example) after vaccination.
* Age > 18 years

Exclusion Criteria:

Group 1 and 2

- Missing informed consent of the subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Toll Like Receptor 7 (TLR7) | Day 1-3 before 1. vaccination
  TLR7 (used method: Whole Genome Sequencing (WGS) using ordinal logistic regression) measured in Single Nucleotide Polymorphism (SNP)
Toll Like Receptor 7 (TLR7) | Day 7-10 after 1. vaccination
  TLR7 (used method: Whole Genome Sequencing (WGS) using ordinal logistic regression) measured in Single Nucleotide Polymorphism (SNP)
Toll Like Receptor 7 (TLR7) | Day 1-3 before 2. vaccination
  TLR7 (used method: Whole Genome Sequencing (WGS) using ordinal logistic regression) measured in Single Nucleotide Polymorphism (SNP)
Toll Like Receptor 7 (TLR7) | Day 7-10 after 2. vaccination
  TLR7 (used method: Whole Genome Sequencing (WGS) using ordinal logistic regression) measured in Single Nucleotide Polymorphism (SNP)
Toll Like Receptor 7 (TLR7) | Month 6-12 after 2. vaccination
  TLR7 (used method: Whole Genome Sequencing (WGS) using ordinal logistic regression) measured in Single Nucleotide Polymorphism (SNP)

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Rieß, Study Director — University Hospital Tübingen
Locations (1):
- University Hospital Tübingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
The COVID19-VAC study will provide data in a pseudonymised manner to national and international databases set up to increase the diagnostic yield through advanced analysis tools and matchmaking against other cohorts
Supporting Information: Analytic Code
Time Frame: Data will become available after analysis and unlimited.